CLINICAL TRIAL: NCT05485415
Title: Personalised Circadian Intervention Study in Elderly With Sleep Problems
Brief Title: Intervention Study in Elderly With Sleep Problems
Acronym: CIEL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mirjam Münch (Network)
Collaborators: University of California (Other)
Responsible Party: Sponsor-Investigator, Mirjam Münch, Principal Investigator, University Psychiatric Clinics Basel
Organization: University Psychiatric Clinics Basel (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-00904
Record Dates: First submitted 2022-06-14; First posted 2022-08-03 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Sleep Disturbance
Keywords: circadian; light; cognition; Zeitgeber; personalized; health; sleep; muliti-modal
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial with a control group
Who Masked: Participant
Masking Description: Participants are unaware whether they are in the intervention or the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Personalised intervention
  Interventions: Behavioral: Multimodal intervention
- Control (Placebo Comparator): General sleep advice
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Multimodal intervention — Participants in the intervention group will receive personalised advice on sleep, light exposure, meal times and physical activity.
  Arms: Intervention
Behavioral: Control — General sleep advice
  Arms: Control

SUMMARY:
The main objective of the study is to improve subjective sleep quality using a multimodal intervention with an intervention and a control group. The multimodal intervention aims to improve circadian Zeitgeber strength. This will be achieved by optimizing daily light exposure, sleep, physical activity, and mealtimes.

DETAILED DESCRIPTION:
The study lasts for 14 months and contains 6 visits. After the screening visit at the Centre for Chronobiology, Basel, Switzerland, participants are assigned to either the intervention or the control group which is followed by a 7-day baseline week at home and a co-design meeting to provide instructions to the intervention and the control group. At the occasion of 2 visits (spread over 6 months) at the participants' homes, different measurements will be performed such as saliva collection, questionnaires, cognitive performance tests, light and rest-activity measures. After the last visit at home, participants come for the second blood sample at the study centre. A follow-up visit 6 months after completion of the last data collection will provide qualitative feedback by the participants.

ELIGIBILITY:
Inclusion Criteria:

at least 65 years old women and men

* Pittsburgh Sleep Quality Index (PSQI) > 5 (indicative of sleep problems)
* Living at home (including self-serviced retirement apartment)

Exclusion Criteria:

* Total blindness or VA < 0.5
* Progressive NCDs (e.g., cancer)
* Acute infections (e.g., Covid-19)
* Neurodegenerative disease
* Psychiatric disease
* Sleep disorder (sleep apnea, narcolepsy)
* Not German speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Subjective sleep quality | 6 months
  Pittsburgh Sleep Quality Index (Score > 5 indicates poor sleep)

SECONDARY OUTCOMES:
Sleep timing | 6 months
  Derived from Activity Watches
Subjective wellbeing | 6 months
  Visual Analogue Scales
Salivary melatonin concentration | 6 months
  Circadian phase marker
Pupil size | 6 months
  Pupil response to chromatic light stimuli
Glucose metabolism | 6 months
  HbA1c concentration (blood)
Telomere length | 6 months
  Age marker
Neuropsychological Battery to assess working memory and attention (including n-back, Psychomotor Vigilance Test) | 6 months
  Cognitive Function

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Münch, PhD, Principal Investigator — Research Associate
Locations (1):
- Centre for Chronobiology, Psychiatric Hopspital of the University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No